CLINICAL TRIAL: NCT03312608
Title: Cerebral Reorganization in Cervical Myelopathy
Brief Title: Cerebral Reorganization in Cervical Myelopathy Measured by Navigated Transcranial Magnetic Stimulation
Acronym: CReMe
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: German Spine Society (Deutsche Wirbelsäulenstiftung) (Other); Insel Gruppe AG, University Hospital Bern (Other); University Hospital of Cologne (Other); University Hospital Munich (Other)
Responsible Party: Principal Investigator, Anna Zdunczyk, principal investigator, physician, Charite University, Berlin, Germany
Other Study IDs: 89830535
Record Dates: First submitted 2017-09-18; First posted 2017-10-18 (Actual); Last update posted 2017-10-18 (Actual); Status verified 2017-10

CONDITIONS: Degenerative Myelopathy
Keywords: cerebral reorganization, TMS

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- mild myelopathy (JOA>12): 40 patients (JOA>12) suffering from symptomatic or asymptomatic degenerative cervical myelopathy scheduled for surgery or conservative treatment. The radiological inclusion criteria are cervical spinal stenosis associated with or without intramedullary high signal intensity lesion on T2-weighted MRI. Exclusion criteria are other pathologies in the vicinity of the corticospinal tract above the lesion site (i.e. tumor, infarction), neuroinflammatory disease, high grade paresis of the upper extremity (BMRC<3), the existence of a cardiac pacemaker, deep brain stimulation electrodes or pregnancy. By means of navigated transcranial magnetic stimulation the resting motor threshold, recruitment curve, cortical silent period and motor area will be determined.
  Interventions: Diagnostic Test: Navigated transcranial magnetic stimulation
- moderate myelopathy: 40 patients (JOA≤12) suffering from symptomatic degenerative cervical myelopathy scheduled for surgery (anterior and/ or posterior decompression) or conservative treatment. The radiological inclusion criteria are cervical spinal stenosis associated with or without intramedullary high signal intensity lesion on T2-weighted MRI. Exclusion criteria are other pathologies in the vicinity of the corticospinal tract above the lesion site (i.e. tumor, infarction), neuroinflammatory disease, high grade paresis of the upper extremity (BMRC<3), the existence of a cardiac pacemaker, deep brain stimulation electrodes or pregnancy. By means of navigated transcranial magnetic stimulation the resting motor threshold, recruitment curve, cortical silent period and motor area will be determined.
  Interventions: Diagnostic Test: Navigated transcranial magnetic stimulation
- healthy control: As a control group, 40 subjects will be included into the study. Exclusion criteria and examination protocol are identical with the patient group. By means of navigated transcranial magnetic stimulation the resting motor threshold, recruitment curve, cortical silent period and motor area will be determined.
  Interventions: Diagnostic Test: Navigated transcranial magnetic stimulation

INTERVENTIONS:
Diagnostic Test: Navigated transcranial magnetic stimulation

SUMMARY:
In degenerative cervical myelopathy (DCM) the dynamics of disease progression and the outcome after surgical decompression vary inter individually and do not necessarily correlate with radiological findings. By better characterization of the underlying pathophysiology this study aims to improve diagnostic power in DCM using Navigated transcranial magnetic stimulation (nTMS).

DETAILED DESCRIPTION:
120 patients with DCM due to cervical spinal canal stenosis will be examined preoperatively and postoperatively with nTMS. On the basis of the initial Japanese Orthopedic Association (JOA) Score two patient groups will be established (JOA≤12/>12). The resting motor threshold, recruitment curve, cortical silent period and motor area will be determined. Accordingly, 40 healthy subjects will be examined.

To the investigators knowledge, this study is the first to analyze changes of corticospinal excitability and reorganization in patients with cervical spondylotic myelopathy with navigated TMS. In the present study, there was a significant difference in parameters of excitability and motor area activation between the severely symptomatic and clinically stable patient group. The investigators analysis showed that chronic CSM induces a recruitment of the non-primary motor area and corticospinal disinhibition, so that axonal damage can be compensated through recruitment of new cortical and supplementary motor connections, to a certain degree. Upon exhaustion of these mechanisms further axonal damage translates directly into new neurological deficits. These results lay the ground for a novel concept in CSM, the "corticospinal reserve capacity".

This study lays the foundation for future research to examine the pathomechanisms in CSM. Functional reorganization occurs on a spinal as well as on a cortical level. The concept of the corticospinal reseve capacity describes a compensatory, increased recruitment of non primary motor areas and corticospinal disinhibition in order to preserve motor function. By detecting the degree of reorganization, a stratification for an unfavourable as well as stable clinical course could be made. This innovative approach to describe the pathomechanisms in CSM might revise current concepts of clinical diagnostics and might have an impact on future treatment strategies.

ELIGIBILITY:
Inclusion Criteria:

* patients with symptomatic/asymptomatic cervical spondylotic myelopathy scheduled for surgery (anterior and/ or posterior decompression) or conservative treatment. The radiological inclusion criteria are cervical spinal stenosis (C3-C7) associated with or without intramedullary high signal intensity lesion on T2-weighted MRI due to disc protrusion or spondylosis.
* healthy subjects without any neurological disease

Exclusion Criteria:

* Exclusion criteria are other pathologies in the vicinity of the corticospinal tract above the lesion site (i.e. tumor, infarction), neuroinflammatory disease, high grade paresis of the upper extremity (BMRC<3), the existence of a cardiac pacemaker, deep brain stimulation electrodes or pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * patients with symptomatic/asymptomatic cervical spondylotic myelopathy scheduled for surgery or conservative Treatment
  * healthy subjects without any neurological disease
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2021-01-01 (Estimated); Study Completion 2023-02-01 (Estimated)

PRIMARY OUTCOMES:
Corticospinal reserve capacity | preoperative
  Comparison of corticospinal reserve capacity (defined by recruitment curve, cortical silent period, motor area) compared to healthy control group
Change in corticospinal reserve capacity | 9 months, 24 months postoperatively
  Postoperative change in corticospinal reserve capacity compared to clinical symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Anna Zdunczyk, M.D., Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Department of neurosurgery Charité, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes
The study results, study protocol and study report will be shared with other Researchers during international congresses and peer reviewed publications
Supporting Information: Study Protocol, SAP, CSR
Time Frame: during the time of the study
Access Criteria: only as a congress presentation or publication presenting the results of the study